CLINICAL TRIAL: NCT06117150
Title: A Pilot Study of the Drug-eluting Coronary Spur StEnt as a Primary trEatment for In-stent Restenosis of the CORONARY Arteries (DEEPER CORONARY)
Brief Title: Pilot Study of the Coronary Spur Stent for In-stent Restenosis (DEEPER CORONARY)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ReFlow Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-008
Record Dates: First submitted 2023-09-28; First posted 2023-11-03 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: In-stent Restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Drug-eluting Coronary Spur StEnt System (Experimental): All subjects enrolled will receive the Drug-eluting Coronary Spur Stent System.
  Interventions: Device: Drug-eluting Coronary Spur Stent System

INTERVENTIONS:
Device: Drug-eluting Coronary Spur Stent System — All subjects enrolled will be treated with the Drug-eluting Coronary Spur Stent System.

SUMMARY:
To demonstrate acceptable short term safety rates of the Drug-eluting Coronary Spur Stent System as a primary treatment for coronary in-stent restenosis.

ELIGIBILITY:
Pre-Procedure Inclusion Criteria:

1. Subject willing and able to provide informed consent and able to comply with the study protocol and follow up. Subjects who are unable to sign due to a physical limitation may have a legal guardian or legally authorized representative (LAR) sign on their behalf.
2. Life expectancy greater than 2 years in the investigator's opinion.
3. Subject is greater than 18 years of age.
4. Female subjects of childbearing potential have a negative pregnancy test ≤ 7 days before the procedure.
5. Endovascular treatment is able to be conducted under non-emergent conditions.
6. Documented stable or unstable angina including non-ST-elevation MI, functional testing demonstrating ischemia, and/or clinical symptoms that in the opinion of the investigator are not amenable to conservative medical therapy and require endovascular intervention.
7. Subject is eligible for dual antiplatelet therapy (DAPT) treatment with aspirin plus P2Y12 inhibitor.

Angiographic Inclusion Criteria:

1. Target vessel is of appropriate size and diameter to be treated with the Coronary Spur Stent.
2. Target lesion is within a previously placed Bare Metal Stent (BMS) or Drug-eluting Stent (DES) and does not extend further than 5mm beyond either the proximal or distal edge of the stent.
3. In-stent restenosis of >50% diameter by angiography.
4. Up to two (2) non-target lesions in non-target vessels may be treated, but successful percutaneous coronary intervention (PCI) of the non-target lesions must be completed before treatment of the target lesion. Successful treatment of a non-target lesion is defined as a residual stenosis of ≤ 30% in 2 near-orthogonal projections with Thrombolysis in Myocardial Infarction (TIMI) 3 flow, as visually assessed by the physician, without the occurrence of prolonged chest pain or ECG changes consistent with MI.
5. Successful pre-dilatation of the target lesion, defined as non-compromised flow or presence of thrombus.

Pre-procedure Exclusion Criteria:

1. Subject unwilling or unlikely to comply with the one-year duration of the study as in the opinion of the investigator.
2. Subject is pregnant, breast-feeding, or is a woman of childbearing potential who is not using appropriate contraceptives.
3. Subject has an active systemic infection that is not controlled at the time of the procedure, including septicemia or bacteremia.
4. Stroke within 90 days of the index procedure.
5. Documented left ventricular ejection fraction (LVEF) <35% by echocardiography.
6. In-stent restenosis occurring in less than 90 days prior to the index procedure.

Impaired renal function (eGFR less than or equal to 25 mL/min) within 30 days of procedure or end stage renal disease on dialysis.

8. History of active peptic ulcer or gastrointestinal bleeding within prior 6 months or other inability to comply with recommended duration of DAPT.

9. Known allergies or sensitivities to heparin, antiplatelet drugs, other anticoagulant therapies which could not be substituted, drug balloon coatings and their excipients, including, but not limited to, paclitaxel, sirolimus, or zotarolimus, or an allergy to contrast media that cannot be adequately pre-treated prior to the index procedure.

10. The subject is currently enrolled in another investigational device or drug trial that interferes with the study endpoints.

11. Known allergy to nitinol or nickel.

12. Any expected elective surgical procedure that would necessitate interruption of DAPT through the 12-month visit.

13. Planned use of atherectomy (rotational, orbital, or laser) device, cutting or scoring balloon.

14. Severe hepatic dysfunction (3 times normal reference values).

15. Planned treatment of additional lesions in target vessel or > two (2) non-target lesions within non-target vessels during index procedure.

16. Target lesion has undergone > two (2) prior stent implant procedures (including the initial index procedure, i.e., > two (2) layers of stent are present at any segment of target lesion).

Angiographic Exclusion Criteria

1. Target lesion is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion.
2. Fractured or otherwise compromised stents in the target vessel or inflow vessel.
3. Target lesion and vessel tortuosity must accommodate the Drug-eluting Coronary Spur.
4. Severe Calcification of the target vessel.
5. Prior history of repeat drug-eluting stent implantation for DES restenosis.
6. Angiographic evidence of thrombus within target artery.
7. Type D dissections or greater incurred during predilitation or crossing (see Appendix II for definitions).
8. Tortuosity of proximal segment or location of In-stent Restenosis (ISR) or extremely angulated segments which prevents tracking of the Coronary Spur Stent to the target lesion.
9. Total occlusions > 3 months old and/or bridging collaterals.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Treatment of the target lesion with the Drug-Eluting Coronary Spur Stent System without occurrence of in-hospital Major Adverse Cardiac Events (MACE). | From time of enrollment procedure through time of post-procedure discharge
  MACE is defined as All-cause death, Myocardial Infarction (MI), any clinically-driven target lesion revascularization (TLR).

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - Auckland City Hospital Te Toka Tumai, Auckland, Grafton
  - Wellington Hospital | Capital, Coast and Hutt Valley, Wellington, Wellington Region

IPD SHARING:
Plan to Share IPD: No